CLINICAL TRIAL: NCT05990595
Title: Evaluation of Health Effects of Adlay on Hyperlipidemia and Hyperglycemia Control (ADL)
Brief Title: Evaluation of Health Effects of Adlay on Hyperlipidemia and Hyperglycemia Control
Acronym: ADL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 202206033RINC
Record Dates: First submitted 2023-07-24; First posted 2023-08-14 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-07

CONDITIONS: Hyperlipidemia; Hyperglycemia; Type 2 Diabetes
Keywords: Adlay, Hyperlipidemia, Hyperglycemia
MeSH Terms: conditions — Hyperlipidemias; Hyperglycemia; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: The clinical trial adopts a randomized cross-over trial, the experimental group to eat white rice with adlay and the control group to eat white rice. Participants in the project were randomly divided into two groups, group A and B, with 30 people in each group. Group A eat 200 gm cooked adlay with white rice to replace their carbohydrates; Group B ate a box of 200 grams of white rice per day. After the first run of study, all participants resume to the original regular diet for two weeks, and then switch groups for crossover trial after the two-week washout period. In the experiment, during the crossover experiment, group A and group B replaced the experimental ingredients, that is, the original white rice group was replaced by adlay with white rice, and the original adlay and white rice group was replaced with white rice for a period of two weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adlay with white rice (Experimental): Group A eat cooked adlay with white rice to replace their carbohydrates: a box of 200 grams of adlay rice per day
  Interventions: Dietary Supplement: Adlay with white rice
- White rice (Placebo Comparator): Group B ate a box of 200 grams of cooked white rice per day
  Interventions: Dietary Supplement: white rice

INTERVENTIONS:
Dietary Supplement: Adlay with white rice — We will investigate the lipid- and glucose-lowering effects of Adlay rice in comparison to white rice through a randomized cross-over trial.
  Arms: Adlay with white rice
Dietary Supplement: white rice — white rice
  Arms: White rice

SUMMARY:
This study explores the efficacy of domestic adlay in improving blood sugar and lipids metabolism, cardiovascular function, and weight control in people with high blood pressure, hyperlipidemia, and hyperglycemia.

Through two weeks of cooked adlay-rice and white rice by a randomized cross-over design to evaluate the lipid- and glucose-lowering effects of adlay on patient with hyperlipidemia and/or hyperglycemia.

DETAILED DESCRIPTION:
Evaluation of health effects of domestic adlay on lowering cholesterol and blood sugar

Hyperlipidemia and diabetes are major risk factors for cardiovascular disease. Clinical experiments have preliminarily proved that phytosterols can help lower blood lipids, and adlay is one of the domestic economic crops that has animal experimental evidence or theoretical potential to be beneficial to blood lipids and blood sugar control, which needs to be further explored and verified. This study explores the efficacy of domestic adlay in improving blood sugar and lipids metabolism, cardiovascular function, and weight control in people with high blood pressure, hyperlipidemia, and hyperglycemia.

We plan to recruit 60 patients with hyperglycemia or hyperlipidemia. aged between 20 and 80 years old, from National Taiwan University Hospital. This study is focused on high blood cholesterol, triglycerides, and hyperglycemia groups, thus participants must have higher cholesterol, triglycerides, or higher fasting blood glucose concentration even under currently stable treatment for at least 6 months. Lipid-lowering and hypoglycemic medication cannot be changed during this trial.

The clinical trial adopts a randomized cross-over trial, the experimental group to eat white rice with adlay and the control group to eat white rice. Participants in the project were randomly divided into two groups, group A and B, with 30 people in each group. Group A eat adlay to replace their carbohydrates: a box of 200 grams of rice (the amount of rice in dry weight is 36 grams of adlay and 54 grams of white rice) per day; Group B ate a box of 200 grams of white rice (the amount of rice was 87 grams based on dry weight) per day. After the first run of study, all participants resume to the original regular diet for two weeks, and then switch groups for crossover trial after the two-week washout period. In the experiment, during the crossover experiment, group A and group B replaced the experimental ingredients, that is, the original white rice group was replaced by adlay with white rice, and the original adlay and white rice group was replaced with white rice for a period of two weeks. To ensure that the test material is homogeneous and uniform, the white rice with adlay is made from the "cooked rice with adlay" produced by Nanqiao Group, HUACIANG INDUSTRY CO., LTD. The adlay cooked rice contains 40% adlay and Taichung No. 194 white rice 60%, and the control group used Taichung No. 194 white rice.

Every participant have to receive blood and urine sampling for biochemical measurement in each stage, 1. Baseline, 2. Two weeks after first stage: adlay with white rice or white rice, 3. Washed period stage for 2 weeks, 4. Two weeks after crossover stage. The main results analysis includes fasting blood sugar,glycosylated hemoglobin, glycosylated hemoglobin, triglycerides, total cholesterol, high-density cholesterol, and low-density cholesterol. Secondary outcome analysis includes blood pressure, body composition analysis, inflammation index, thyroid function, levels of intestinal hormones (cholecystokinin, gastrin) and glucagon-like peptide-1, and other emerging blood lipid indicators, such as small-dense LDL-C. The above measurements will be performed every 2 weeks for each stage. Pittsburgh Sleep Quality Index and Center for Epidemiological Studies Depression Scale (CES-D) will also be assessed every 2 weeks for each stage.

Keywords: hyperlipidemia, hyperglycemia, diabetes mellitus, randomized crossover trial

ELIGIBILITY:
Inclusion Criteria:

1. Hyperlipidemia: Levels of LDL-choleterol equal or greater than 130 mg/dL, or triglyceride equal or greater than 150 mg/dL
2. Hyperglycemia: fasting glucose equal or greater than 100 mg/dL

Exclusion Criteria:

Secondary hyperglycemia Secondary hyperlipidemia

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-07-07 (Actual); Primary Completion 2023-09-28 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Fasting blood glucose | 2 weeks for each stage
  glucose-lowering effects
Cholesterol | 2 weeks for each stage
  Lipids
HDL-cholesterol | 2 weeks for each stage
  Lipids
LDL-cholesterol | 2 weeks for each stage
  Lipids
Triglycerides | 2 weeks for each stage
  Lipids
Glycosylated hemoglobin (HbA1C) | 2 weeks for each stage
  Hemoglobin A1C is a form of hemoglobin (Hb) that is chemically linked to sugar

SECONDARY OUTCOMES:
Blood pressure | 2 weeks for each stage
  physiological biomarkers
Body composition | 2 weeks for each stage
  The percentages of fat, bone and muscle in human bodies by bioelectric impedance technology
hs-CRP (high sensitivity C-reactive protein) | 2 weeks for each stage
  Inflammation
Free T4 and TSH (Thyroid Stimulating Hormone) | 2 weeks for each stage
  Thyroid function tests
Insulin | 2 weeks for each stage
  A peptide hormone produced by beta cells of the pancreatic islets
Gastrin, Cholecystokinine, and Glucagon-like peptide 1 | 2 weeks for each stage
  Intestin Hormones
Small-dense LDL-cholesterol | 2 weeks for each stage
  LDL subpopulation particles

OTHER OUTCOMES:
Pittsburgh Sleep Quality Index | 2 weeks for each stage
  Sleep quality assessment
Center for Epidemiologic Studies Depression Scale (CES-D), NIMH | 2 weeks for each stage
  Depression scale assessment

CONTACTS AND LOCATIONS:
Overall Officials: Ta-Chen Su, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan